CLINICAL TRIAL: NCT02495311
Title: The Association Between Adenomyosis/Uterine Myoma and Lower Urinary Tract Symptoms and Gastrointestinal Symptoms
Brief Title: The Association Between Adenomyosis/Uterine Myoma and Lower Urinary Tract Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 103129-F
Record Dates: First submitted 2015-07-04; First posted 2015-07-13 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Adenomyosis; Uterine Leiomyoma
Keywords: adenomyosis; uterine myoma; lower urinary tract symptoms; sexual dysfunction; gastrointestinal symptom
MeSH Terms: conditions — Adenomyosis; Myofibroma; Lower Urinary Tract Symptoms; Sexual Dysfunction, Physiological | interventions — Uterine Myomectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Women with uterine myoma: Women with uterine myoma
  Interventions: Procedure: myomectomy or adenomyomectomy
- Women with adenomyosis: Women with adenomyosis
  Interventions: Procedure: myomectomy or adenomyomectomy
- Women without uterine myoma or adenomyosis: Control group

INTERVENTIONS:
Procedure: myomectomy or adenomyomectomy
  Groups: Women with adenomyosis; Women with uterine myoma

SUMMARY:
The aim of this study is to assess the relationship between adenomyosis/myoma and lower urinary tract symptoms, sexual function and gastrointestinal symptoms.

DETAILED DESCRIPTION:
All outpatient patients were found to have >3 cm uterine myoma or adenomyosis were invited to participate in this study. The size and location of uterine myoma or adenomyosis and the uterus should be assessed by ultrasonography. Besides, all enrolled female patients will be asked to complete overactive bladder symptom score, female bladder function (UDI-6 & IIQ-7), female sexual function index, and bowel incontinence assessment questionnaires. In addition, patients who underwent surgeries for myoma or adenomyosis will be requested to complete the above questionnaires at 3 months after surgery. Women with intact uterus should be assessed again by ultrasonography. At least 30 women with age and body mass index matched and without uterine myoma or adenomyosis will be invited to participate in this study as the control group.

ELIGIBILITY:
<Women with myoma or adenomyosis>

Inclusion Criteria:

1. >20 years old.
2. Myoma: women with >3 cm uterine myoma
3. Adenomyosis: women with uterus having several dark area (lacunar areas) in one uterine wall or thickening uterine wall

<The control group>

Inclusion criteria:

1. >20 years old.
2. Women without myoma or adenomyosis

<Both groups>

Exclusion Criteria:

1. The patient has a lower urinary tract infection or acute intestinal inflammation.
2. Previous surgery for the bladder or urethra.
3. History of urinary tract stones or tumors.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with uterine myoma or adenomyosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-11-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The corrleation coefficient between the size of myoma and Overactive Bladder Symptoms Scores | 12 weeks
  The Spearman's correlation between the size of uterine myoma and the score of Overactive Bladder Symptoms Scores

SECONDARY OUTCOMES:
The corrleation coefficient between the size of myoma and the presence of constipation/diarrhea | 12 weeks
  The Spearman's correlation between the size of uterine myoma and the presence of constipation/diarrhea
Comparison of Overactive Bladder Symptoms Scores between the adenomyosis group and the control group | 12 weeks
  Comparison of Overactive Bladder Symptoms Scores between the adenomyosis group and the control group by Wilcoxon rank-sum test
Comparisons of the constipation/diarrhea rates between the adenomyosis group and the control group | 12 weeks
  Comparisons of the constipation/diarrhea rates between the adenomyosis group and the control group by Chi-square test or Fisher's exact test

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital, Banqiao, New Taipei, Taiwan
Locations (1):
- Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan